CLINICAL TRIAL: NCT00838383
Title: SELECTIVE ENDOTHELIN TYPE A RECEPTOR INHIBITION IN CARDIAC SURGERY SUBJECTS WITH PRE-EXISTING CARDIOVASCULAR RISK FACTORS: A DOSE CONFIRMATION STUDY
Brief Title: Confirming The Sitaxsentan Dose In Patients Undergoing Heart Surgery
Acronym: FCAD02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1321004; B1321004; FCAD02-CARDIAC SURGERY (Other: Alias Study Number)
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Surgery Subjects; Subjects Undergoing CABG and/or Cardiac Valve Replacement
Keywords: multi-center; placebo-controlled; randomized study of sitaxsentan administered to subjects post-cross-clamp release and 12 hours post-CPB
MeSH Terms: interventions — sitaxsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- sitaxsentan (1.0 mg/kg) (Experimental)
  Interventions: Drug: sitaxsentan (Thelin)
- sitaxsentan (2.0 mg/kg) (Experimental)
  Interventions: Drug: sitaxsentan (Thelin)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sitaxsentan (Thelin) — sitaxsentan (1.0 mg/kg) will begin immediately following cross-clamp release and 12 hours post-CPB.
  Other Names: sitaxsentan, Thelin
  Arms: sitaxsentan (1.0 mg/kg)
Drug: sitaxsentan (Thelin) — Sitaxsentan (2.0 mg/kg) will begin immediately following cross-clamp release and 12 hours post-CPB.
  Other Names: sitaxsentan, Thelin
  Arms: sitaxsentan (2.0 mg/kg)
Drug: Placebo — Placebo will begin immediately following cross-clamp release and 12 hours post-CPB.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized study of sitaxsentan administered intravenously to subjects who are undergoing elective CABG, cardiac valve replacement, or combined CABG and cardiac valve replacement procedures that require CPB.

ELIGIBILITY:
Inclusion Criteria:

* Has been identified for coronary artery bypass grafting (CABG), aortic and/or mitral valve replacement, or combined CABG and cardiac valve replacement procedures that require cardiopulmonary bypass (CPB).

Exclusion Criteria:

* Requires an emergent or "emergency" CABG and/or cardiac valve replacement.

Ages: 48 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-08-10 (Actual); Primary Completion 2008-03-31 (Actual); Study Completion 2008-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Pennsylvania,, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Chattanooga Heart Institute, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321004&StudyName=Confirming%20The%20Sitaxsentan%20Dose%20In%20Patients%20Undergoing%20Heart%20Surgery

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitaxsentan (1 mg/kg): Participants received single intravenous (IV) infusion of sitaxsentan 1 milligram per kilogram (mg/kg) immediately following cross-clamp release and at 12 hours post-cardiopulmonary bypass (CPB).
- Sitaxsentan (2 mg/kg): Participants received single IV infusion of sitaxsentan 2 mg/kg immediately following cross-clamp release and at 12 hours post-CPB.
- Placebo: Participants received placebo (matched to sitaxsentan) immediately following cross-clamp release and at 12 hours post-CPB.
Period: Overall Study
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Started | 9 | 10 | 10
Completed | 9 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received either sitaxsentan 1 mg/kg, sitaxsentan 2 mg/kg, or placebo during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.86) | 68.5 (8.81) | 67.2 (6.56) | 66.1 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 7 | 10 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From 0 Hour in Pulmonary Vascular Resistance (PVR) at 0.5 Hour Post-separation From Cardiopulmonary Bypass (CPB)
Description: PVR in participants was derived from mean pulmonary artery pressure (PAP) (millimeter of mercury [mmHg]), pulmonary capillary wedge pressure (PCWP [mmHg]) and cardiac output (CO [litres per minute]). It was calculated using the following formula: ([mean PAP-PCWP] divided by CO)*80, where CO= stroke volume (SV)*heart rate (HR). Post-separation from CPB was the time immediately following cross-clamp release in CPB. Percent change in PVR at 0.5 hour post-separation from CPB in participants were summarized and reported.
Time Frame: 0 hour, 0.5 hour post-separation from CPB
Population: Safety analysis set included all participants who received either sitaxsentan 1 mg/kg, sitaxsentan 2 mg/kg, or placebo during the study. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 9 | 10
percent change | -7.75 (55.277) | -10.94 (37.967) | 62.22 (260.172)
Statistical Analysis 1: Comparison: Sitaxsentan (1 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.5307, ANCOVA; Mean Difference (Net) = -70.0, 95% CI 2-sided [-291.3 to 151.4]
Statistical Analysis 2: Comparison: Sitaxsentan (2 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.5121, ANCOVA; Mean Difference (Net) = -73.2, 95% CI 2-sided [-294.5 to 148.2]

2. Primary Outcome: Percent Change From 0 Hour in Pulmonary Vascular Resistance (PVR) at 6 Hour Post-separation From Cardiopulmonary Bypass (CPB)
Description: PVR in participants was derived from mean PAP (mmHg), PCWP (mmHg) and CO (litres per minute). It was calculated using the following formula: ([mean PAP-PCWP] divided by CO)*80, where CO= SV * HR. Percent change in PVR at 6 hour in participants were summarized and reported.
Time Frame: 0 hour, 6 hour post-separation from CPB
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 9 | 9
percent change | 39.36 (61.615) | -12.01 (39.561) | 173.68 (511.269)
Statistical Analysis 1: Comparison: Sitaxsentan (1 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.2735, ANCOVA; Mean Difference (Net) = -123.1, 95% CI 2-sided [-345.5 to 99.3]
Statistical Analysis 2: Comparison: Sitaxsentan (2 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.1223, ANCOVA; Mean Difference (Net) = -174.5, 95% CI 2-sided [-396.8 to 47.9]

3. Primary Outcome: Percent Change From 0 Hour in Pulmonary Vascular Resistance (PVR) at 12 Hour Post-separation From Cardiopulmonary Bypass (CPB)
Description: PVR in participants was derived from mean PAP (mmHg), PCWP (mmHg) and CO (litres per minute). It was calculated using the following formula: ([mean PAP-PCWP] divided by CO)*80, where CO= SV * HR. Percent change in PVR at 12 hour in participants were summarized and reported.
Time Frame: 0 hour, 12 hour post-separation from CPB
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 9 | 10
percent change | 31.42 (67.887) | -12.32 (37.517) | 98.03 (283.333)
Statistical Analysis 1: Comparison: Sitaxsentan (1 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.5505, ANCOVA; Mean Difference (Net) = -66.6, 95% CI 2-sided [-288.0 to 154.8]
Statistical Analysis 2: Comparison: Sitaxsentan (2 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.3237, ANCOVA; Mean Difference (Net) = -110.3, 95% CI 2-sided [-331.7 to 111.0]

4. Primary Outcome: Percent Change From 0 Hour in Pulmonary Vascular Resistance (PVR) at 24 Hour Post-separation From Cardiopulmonary Bypass (CPB)
Description: PVR in participants was derived from mean PAP (mmHg), PCWP (mmHg) and CO (litres per minute). It was calculated using the following formula: ([mean PAP-PCWP] divided by CO)*80, where CO= SV * HR. Percent change in PVR at 24 hour in participants were summarized and reported.
Time Frame: 0 hour, 24 hour post-separation from CPB
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 8 | 9
percent change | 18.06 (63.362) | -15.99 (41.604) | 195.64 (522.379)
Statistical Analysis 1: Comparison: Sitaxsentan (1 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.1412, ANCOVA; Mean Difference (Net) = -166.5, 95% CI 2-sided [-389.6 to 56.6]
Statistical Analysis 2: Comparison: Sitaxsentan (2 mg/kg) vs Placebo; Test type: Superiority or Other; p = 0.0813, ANCOVA; Mean Difference (Net) = -199.8, 95% CI 2-sided [-425.0 to 25.5]

5. Primary Outcome: Mortality: Number of Participants Died During Surgery and Initial Hospitalization
Description: Number of participants who died during surgery or during initial hospitalization are reported here.
Time Frame: During surgery, initial hospitalization period (up to 29 days for 1 mg/kg group, up to 44 days for 2 mg/kg dose group, up to 19 days for placebo group)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
participants
  During surgery | 0 | 0 | 0
  During initial hospitalization | 2 | 1 | 0

6. Primary Outcome: Number of Participants With Myocardial Infarction, Cerebrovascular Event, Hemodynamic Collapse and Re-operation
Description: Number of participants with following incidents: myocardial infarction (Q and non-Q wave); stroke or cerebrovascular event (acute ischemia, hemorrhagic stroke or infarction, or a transient ischemia attack); hemodynamic collapse (requiring ventricular assistance devices) and re-operation (participants who returned to the operating room) during the initial hospitalization were reported.
Time Frame: Initial hospitalization period (up to 44 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
participants
  Myocardial Infarction | 1 | 0 | 0
  Stroke or Cerebrovascular event | 0 | 0 | 0
  Hemodynamic collapse | 1 | 2 | 0
  Re-operation | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Inotropic Requirements During the 24 Hours Postoperative Period
Description: Participants were considered for inotropic requirements/therapy in case of either severe right ventricular failure or high pulmonary artery pressure, or if cardiac output was not maintained with epinephrine.
Time Frame: Immediately after cross-clamp removal up to 24 hours post-separation from CPB
Population: Data was not collected, since this outcome was not analyzed as per Sponsor's discretion.
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From 0 Hour in Cardiac Output (CO) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: CO was calculated by multiplying stroke volume (SV) with heart rate (HR). It was used to evaluate the hemodynamic profile of each participant.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: Safety analysis set included all participants who received either sitaxsentan 1 mg/kg, sitaxsentan 2 mg/kg, or placebo during the study. Missing values were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
liters per minute
  At 0 hour post-separation from CPB | 5.48 (2.036) | 5.51 (1.211) | 4.83 (1.158)
  Change at 0.5 hours post-separation from CPB | 0.22 (0.696) | -0.36 (0.973) | 0.16 (0.532)
  Change at 6 hours post-separation from CPB | 0.38 (2.138) | 0.61 (2.088) | 0.43 (1.299)
  Change at 12 hours post-separation from CPB | 1.32 (1.552) | 0.00 (1.505) | 0.52 (1.045)
  Change at 24 hours post-separation from CPB | 1.40 (2.636) | 0.21 (1.782) | 0.48 (1.403)

9. Secondary Outcome: Change From 0 Hour in Central Venous Pressure (CVP) at 0.5, 6, 12, and 24 Hours Post-separation From Cardiopulmonary Bypass (CPB)
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: Safety analysis set included all participants who received either sitaxsentan 1 mg/kg, sitaxsentan 2 mg/kg, or placebo during the study. Missing values were imputed using the LOCF method. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 9
millimeters of mercury (mmHg)
  At 0 hour post-separation from CPB | 9.89 (8.724) | 8.10 (5.425) | 9.22 (5.518)
  Change at 0.5 hours post-separation from CPB | 2.11 (2.804) | 0.40 (1.578) | 0.33 (4.301)
  Change at 6 hours post-separation from CPB | 0.78 (10.146) | 5.70 (6.750) | 1.44 (6.540)
  Change at 12 hours post-separation from CPB | 0.00 (9.220) | 3.80 (5.846) | 3.11 (7.044)
  Change at 24 hours post-separation from CPB | 1.89 (9.649) | 3.90 (6.740) | 0.78 (7.311)

10. Secondary Outcome: Change From 0 Hour in Hematocrit at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: The hematocrit is percentage of the volume of whole blood that is made up of red blood cells (RBCs).
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: Safety analysis set included all participants who received either sitaxsentan 1 mg/kg, sitaxsentan 2 mg/kg, or placebo during the study. Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
percentage of red blood cells in blood
  0 hour post-separation from CPB | 25.56 (4.157) | 26.46 (1.984) | 25.30 (2.541)
  Change at 0.5 hours post-separation from CPB | 1.77 (2.422) | 3.29 (2.804) | 2.30 (2.541)
  Change at 6 hours post-separation from CPB | 9.64 (4.081) | 6.82 (5.310) | 7.55 (5.204)
  Change at 12 hours post-separation from CPB | 8.93 (4.013) | 5.52 (3.862) | 7.68 (4.757)
  Change at 24 hours post-separation from CPB | 7.07 (4.060) | 5.77 (4.098) | 8.25 (3.925)

11. Secondary Outcome: Change From 0 Hour in Heart Rate at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: Heart rate was assessed as one of the hemodynamic profile assessments at the specified time points.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
beats per minute (bpm)
  0 hour post-separation from CPB | 80.11 (13.851) | 84.50 (16.298) | 77.80 (9.102)
  Change at 0.5 hours post-separation from CPB | -1.56 (9.580) | -1.70 (11.225) | -2.80 (8.351)
  Change at 6 hours post-separation from CPB | 5.00 (21.593) | 1.10 (16.980) | -2.00 (11.804)
  Change at 12 hours post-separation from CPB | 8.11 (12.098) | 0.00 (18.868) | 0.70 (21.474)
  Change at 24 hours post-separation from CPB | 11.56 (17.350) | 1.40 (13.074) | 0.80 (18.408)

12. Secondary Outcome: Change From 0 Hour in Mean Pulmonary Artery Pressure (MPAP) at 0.5, 6, 12, and 24 Hours Post-separation From Cardiopulmonary Bypass (CPB)
Description: mPAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position. It was used to evaluate the hemodynamic profile of each participant.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
mmHg
  At 0 Hour post-separation from CPB | 19.27 (7.224) | 26.02 (10.392) | 20.81 (6.978)
  Change at 0.5 hours post-separation from CPB | -1.14 (4.765) | -3.51 (7.321) | -0.41 (6.276)
  Change at 6 hours post-separation from CPB | 3.12 (7.576) | 2.41 (7.834) | 2.41 (9.676)
  Change at 12 hours post-separation from CPB | 2.88 (6.468) | 0.41 (8.832) | 3.80 (7.246)
  Change at 24 hours post-separation from CPB | 4.92 (7.253) | 0.22 (10.727) | 1.96 (9.046)

13. Secondary Outcome: Change From 0 Hour in Pulmonary Capillary Wedge Pressure (PCWP) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure. It was used to evaluate the hemodynamic profile of each participant.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 8 | 7 | 8
mmHg
  0 Hour post-separation from CPB | 10.38 (7.652) | 14.43 (4.962) | 12.50 (5.292)
  Change at 0.5 hours post-separation from CPB | 0.25 (3.694) | -0.43 (1.618) | -0.88 (2.232)
  Change at 6 hours post-separation from CPB | 0.38 (6.823) | 2.71 (4.152) | -0.63 (4.868)
  Change at 12 hours post-separation from CPB | -0.75 (7.005) | 3.57 (4.826) | 0.00 (6.949)
  Change at 24 hours post-separation from CPB | -0.25 (7.265) | 2.86 (5.146) | -2.25 (6.519)

14. Secondary Outcome: Change From 0 Hour in Pulmonary Vascular Resistance (PVR) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: PVR in participants was derived from mean PAP (mmHg), PCWP (mmHg) and CO (litres per minute). It was calculated using the following formula: ([mean PAP-PCWP] divided by CO)*80, where CO= SV * HR.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: (dynes*second) per centimeter^5
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 9
(dynes*second) per centimeter^5
  At 0 Hour post-separation from CPB | 125.28 (74.325) | 166.22 (81.090) | 112.79 (59.363)
  Change at 0.5 hours post-separation from CPB | -31.32 (71.465) | -33.47 (94.027) | -4.04 (52.134)
  Change at 6 hours post-separation from CPB | 19.31 (66.920) | -33.53 (95.697) | 33.99 (89.573)
  Change at 12 hours post-separation from CPB | 7.40 (58.674) | -29.66 (98.021) | 28.49 (58.749)
  Change at 24 hours post-separation from CPB | 0.21 (68.221) | -33.60 (87.893) | 55.33 (80.563)

15. Secondary Outcome: Change From 0 Hour in Venous Oxygen Saturation (SV02/02) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: Venous oxygen saturation is the percentage of oxygen bound to hemoglobin in blood returning to the right side of the heart. It reflects the amount of oxygen "left over" after the tissues consumption.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 7 | 8 | 9
percentage of oxygen saturation
  At 0 hour post-separation from CPB | 75.14 (14.949) | 73.25 (10.053) | 72.44 (22.305)
  Change at 0.5 hours post-separation from CPB | 0.14 (6.644) | 0.88 (4.086) | 2.44 (7.055)
  Change at 6 hours post-separation from CPB | -4.29 (12.459) | -8.50 (7.191) | -0.44 (8.719)
  Change at 12 hours post-separation from CPB | -3.00 (11.328) | -8.75 (4.803) | -1.22 (8.059)
  Change at 24 hours post-separation from CPB | -5.14 (11.006) | -14.38 (9.591) | -0.78 (6.815)

16. Secondary Outcome: Change From 0 Hour in Systemic Vascular Resistance (SVR) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Description: SVR was calculated using formula: ([mean systemic arterial pressure - mean right atrial pressure] divided by CO)*80, where CO= SV * HR.
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: (dynes*second) per centimeter^5
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
(dynes*second) per centimeter^5
  At 0 hour post-separation from CPB | 978.37 (490.306) | 959.89 (281.280) | 1155.39 (521.235)
  Change at 0.5 hours post-separation from CPB | -117.39 (229.848) | 1.14 (214.493) | -20.25 (255.252)
  Change at 6 hours post-separation from CPB | 89.96 (511.943) | -139.23 (330.787) | -77.92 (673.047)
  Change at 12 hours post-separation from CPB | -216.84 (407.566) | -63.12 (343.174) | -193.43 (562.028)
  Change at 24 hours post-separation from CPB | -80.49 (358.157) | 26.74 (384.919) | -8.37 (663.864)

17. Secondary Outcome: Change From 0 Hour in Mean Systemic Blood Pressure (MSBP) at 0.5, 6, 12, and 24 Hours Post-Separation From Cardiopulmonary Bypass (CPB)
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
mmHg
  At 0 hour post-separation from CPB | 69.01 (13.887) | 71.90 (12.768) | 72.55 (11.760)
  Change at 0.5 hours post-separation from CPB | -5.80 (15.467) | -3.70 (11.658) | 2.21 (13.509)
  Change at 6 hours post-separation from CPB | 6.30 (15.133) | 1.97 (12.846) | 3.04 (14.554)
  Change at 12 hours post-separation from CPB | 1.15 (15.240) | 0.73 (11.124) | 0.39 (17.768)
  Change at 24 hours post-separation from CPB | 11.93 (13.039) | 8.20 (14.764) | 8.00 (20.338)

18. Secondary Outcome: Change From 0 Hour in Urine Output at 0.5, 6, 12, and 24 Hours Post-separation From Cardiopulmonary Bypass (CPB)
Time Frame: 0, 0.5, 6, 12, 24 hours post-separation from CPB
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 8
milliliters (mL)
  At 0 hour post-separation from CPB | 105.56 (196.365) | 124.50 (162.830) | 107.50 (117.959)
  Change at 0.5 hours post-separation from CPB | -42.11 (186.162) | 0.50 (136.472) | -16.88 (185.817)
  Change at 6 hours post-separation from CPB | 664.78 (657.273) | 334.50 (325.358) | 367.50 (546.083)
  Change at 12 hours post-separation from CPB | 520.78 (637.651) | 358.00 (485.038) | 145.63 (244.298)
  Change at 24 hours post-separation from CPB | 611.78 (785.270) | 579.80 (641.390) | 443.75 (790.672)

19. Secondary Outcome: Number of Participants With Unanticipated Perioperative and Postoperative Blood Requirements
Description: Number of participants with unanticipated perioperative (occurring at or around the time of the surgery) and postoperative (period following the surgery) blood requirements were recorded on case report forms, summarized and reported in this outcome measure.
Time Frame: 0 to 24 hours post-separation from CPB
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
participants | 0 | 3 | 0

20. Secondary Outcome: Duration of Assisted Ventilation
Description: Assisted Ventilation time was the time (in hours) between intubation and extubation.
Time Frame: 0 hour up to 24 hours post-separation from CPB
Population: as for baseline characteristics
Measure: Median (Full Range); unit: hours
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
hours | 12 (23.2) [9 to 72] | 23 (39.7) [9 to 143] | 21 (10.6) [10 to 47]

21. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Time Frame: 0 hour post-separation from CPB up to 44 days
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
days | 4 (2.5) [2 to 10] | 6 (10.7) [3 to 37] | 5 (2.1) [4 to 10]

22. Secondary Outcome: Duration of Initial Postoperative Hospitalization
Description: The duration of initial postoperative hospitalization had been reported.
Time Frame: 0 hour post-separation from CPB up to 44 days
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Number analyzed (Participants) | 9 | 10 | 10
days | 8 (8.2) [4 to 29] | 11 (13.5) [5 to 44] | 10 (3.9) [6 to 19]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan (1 mg/kg) | Sitaxsentan (2 mg/kg) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/9 | 5/10 | 4/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (1 mg/kg) (N=9) | Sitaxsentan (2 mg/kg) (N=10) | Placebo (N=10)
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (1 mg/kg) (N=9) | Sitaxsentan (2 mg/kg) (N=10) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 5 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Vascular resistance systemic decreased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 3 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 2
Thrombosis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.